CLINICAL TRIAL: NCT03593109
Title: A Single-center Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LCAR-L10D Cell Formulations Targeting CD19 and CD22 in Patients With CD19- and/or CD22-Positive Relapsed/Refractory B-cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Suitable patients were not recruited
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Legend-CART-201803-Ⅱ
Record Dates: First submitted 2018-07-07; First posted 2018-07-19 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma, B-Cell
Keywords: Chimeric Antigen Receptor T cells; CD19 and CD22
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-L10D treatment group (Experimental): In LCAR-L10D treatment group, patients will be treated with dual specificity CD19 and CD22 CAR-T cells with a escalation approach, 3 CAR-T dosage will be tested in this study: 0.5×10^6, 1.5×10^6, 5.0×10^6 CAR-T cells/kg.
  Interventions: Drug: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy

INTERVENTIONS:
Drug: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy — Patients will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of CAR-T cells. After a pre-treatment lymphodepletion therapy, patients will receive the Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy by intravenous injection.

SUMMARY:
This is a prospective, single-arm, single-center, open-label, single-dose dose finding and expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy profile of LCAR-L10D in subjects with CD19- and/or CD22-positive relapsed/refractory B-cell lymphoma after prior adequate standard of care.

DETAILED DESCRIPTION:
CD19-directed CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory B-cell malignancies, CD19 and CD22 are proteins usually expressed on the surface of the lymphoma cells. The dual specificity CAR enables the T-cells to recognize and kill the tumor cell through recognition of CD19 and CD22.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical study; fully understand and be informed of the information on this study, and sign the written Informed Consent Form (ICF); willing to follow and able to complete all trial procedures.
2. According to the criteria for B-cell lymphoma defined in the National Comprehensive Cancer Network (NCCN) Guidelines for Lymphoma (5th edition 2018), and with CD19- and/or CD22-positive lymphoma cells detected by flow cytometry or immunohistochemistry;
3. Must have at least 1 evaluable or measurable lesion meeting Lugano 2014 criteria [Evaluable lesions: Fluorodeoxyglucose/positron emission tomography (FDG/PET) showed increased local uptake in lymph nodes or extranodal sites (higher than the liver), and PET and/or computed tomography (CT) findings are consistent with lymphoma manifestations. Measurable lesions: defined as nodule lesions with a long diameter greater than 15 or extranodal lesions with a long diameter greater than 10 mm (if the only measurable lesion has been previously treated with radiation therapy, the evidence of radiographic progression after radiation therapy is required), with increased FDG uptake). Absence of measurable lesion and diffuse increase of hepatic FDG uptake should be excluded.
4. Relapsed/refractory BCL (meet one of the following conditions):

   1. Subjects in this category had received at least two cycles of two or more lines of standard of care and had been evaluated for best clinical response per Lugano 2014 at the time of enrollment: (one of the following conditions are met)

      * The subject had a best clinical response of PD after the most recent standard chemotherapy;
      * The subject had a best clinical response of SD after the most recent standard chemotherapy, but PD occurred when SD persisted for less than 6 months;
   2. Recurrence or progression within ≤ 12 months after autologous hematopoietic stem cell transplantation;
   3. In one of the following situations, the benefit of the subject may outweigh the risk as judged jointly by the investigator and the partner:

      * The subject had received at least two lines of standard of care, and the best response after the most recent standard chemotherapy was SD, which persisted for less than 6 months, and the evaluable or measurable disease was larger than before but did not achieve PD;
      * The subject had received at least two lines of standard of care, and the best response after the most recent standard chemotherapy was partial response (PR) or higher, but persisted for less than 6 months before progression;
      * The subject had received at least two lines of standard of care and was intolerant to the most recent chemotherapy.
5. All subjects must have received standardized treatment regimens with anti-CD20 monoclonal antibodies (except for those with CD20-negative tumors as determined by the investigator) and anthracyclines. For standardized treatment regimens, please refer to the criteria in the NCCN Guidelines for B-cell Lymphoma (version 5, 2018);
6. Male or female, aged 18-75 years at the time of signing the ICF;
7. Primary laboratory test values met the following criteria to demonstrate adequate organ and bone marrow function without severe hematopoietic abnormalities and heart, lung, liver, renal dysfunction and immunodeficiency:

   Serum albumin ≥30g/L Haemoglobin ≥ 8.0 g/dL (no red blood cell [RBC] infusion within 7 days prior to laboratory tests; recombinant human erythropoietin is allowed) * Absolute neutrophil count ≥ 0.75 × 109/L (growth factor support is allowed but must not have received supportive care within 7 days prior to laboratory tests) Platelet ≥ 40 × 109/L (must not have received blood transfusion support within 7 days prior to laboratory tests) Creatinine clearance ≥ 40 mL/min/1.73 m2, calculated according to Modified Dietary Formula for Renal Disease (Attachment 11) or 24-hour urine collection results.

   ALT and AST ≤ 3.0 x upper limit of normal (ULN) Total bilirubin ≤ 2.0 × ULN; except for subjects with congenital bilirubinemia, such as Gilbert's syndrome (in this case, direct bilirubin ≤ 1.5 x ULN is required) Coagulation PT and APTT <2ULN SpO2 ≥95%

   * For subjects who meet the inclusion criteria at screening, red blood cell infusion after the first hematology test at screening is allowed to maintain hemoglobin levels ≥ 8.0 g/dL.
8. ECOG performance status of 0-1;
9. Estimated survival time of patients > 90 days;
10. A highly sensitive serum pregnancy test (beta human chorionic gonadotropin [beta-HCG]) must be negative at screening and prior to first treatment with cyclophosphamide and fludarabine in women of childbearing potential.
11. Women of childbearing potential must comply with the following requirements:

    * Subjects must agree to use a highly effective method of contraception (annual failure rate < 1% for continuous and correct use) and agree to use a highly effective method of contraception from signing the informed consent form (ICF) until at least 1 year after receiving infusion of LCAR-L10D cell formulation. Highly effective methods of contraception include:

      * User-independent methods: 1) implantable progesterone contraceptives that inhibit ovulation; 2) intra-uterine devices (IUDs); intrauterine hormone-releasing systems; 3) vasectomies in sexual partners;
      * User-dependent methods: 1) compound (estrogen- and progestogen-containing) hormonal contraceptives that inhibit ovulation: oral, vaginal and transdermal; 2) progesterone contraceptives (oral or injectable) that inhibit ovulation.

In addition to highly effective methods of contraception, male subjects should:

* Agree to use barrier contraception (e.g. condoms plus spermicidal foam/gel/film/emulsion/suppository) upon sexual intercourse with a woman of childbearing potential from signing the ICF to at least 1 year after receiving infusion of the LCAR-L10D cell formulation.
* Use condoms when having sex with a pregnant woman Women and men must agree not to donate ova (oocytes, oocytes) or sperm during the study and within 1 year after infusion of LCAR-L10D cell formulation.

Note: Hormonal contraceptives may interact with study treatment, resulting in decreased contraceptive efficacy.

Exclusion Criteria:

1. Subjects who have received any CART cell therapy or other genetically modified T cell therapy;
2. Previous allogeneic stem cell transplantation.
3. Have been diagnosed or treated with other aggressive malignancies other than B-cell lymphoma, with the following exceptions:

   1. Malignant tumors that have been treated radically, and no known active disease within ≥ 2 years prior to enrollment; or
   2. Non-melanoma skin cancers have been adequately treated without symptom of disease.
4. Previous anti-tumor therapy (prior to apheresis) as follows:

   1. Targeted therapy, epigenetic therapy, or investigational drug within 14 days or at least 5 half-lives (whichever is shorter), or has used an invasive investigational medical device.
   2. Cytotoxic drugs within 14 days.
   3. Immunomodulator within 7 days.
   4. Monoclonal antibodies to treat BCL within 21 days.
   5. Radiation therapy within 14 days.
5. Positive for any one of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus antibody (HIV-Ab)
6. The following cardiac disorders occurred:

   1. New York Heart Association (NYHA) phase III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) ≤ 6 months prior to enrollment;
   3. History of clinically significant ventricular arrhythmia or unexplained syncope (non-vasovagal or caused by dehydration);
   4. History of severe nonischemic cardiomyopathy;
   5. Impaired cardiac function (LVEF < 50%) as assessed by echocardiogram or multiple gated acquisition scan (MUGA) (performed ≤ 8 weeks prior to apheresis).
   6. Clinically significant pericardial effusion
7. Clinically significant pleural effusion（Excluding caused by lymphoma mass compression or pleural involvement）;
8. Except alopecia or peripheral neuropathy, other toxicity of prior anti-tumor therapy must have improved to baseline or ≤ Grade 1.
9. Patients with serious underlying diseases, such as:

   1. Documented serious active viral or bacterial infection, or uncontrolled systemic fungal infections;
   2. Active auto-immune diseases or medical history of auto-immune diseases within 3 years;
   3. Clear clinical evidence of dementia or altered mental status.
10. Female subjects who become pregnant, are breastfeeding, or plan to become pregnant while participating in the study or within 1 year after receiving study treatment;
11. Male subjects who plan to have a baby while participating in the study or within 1 year after receiving study treatment;
12. Subjects with marked bleeding tendency, e.g, digestive tract hemorrhage, coagulation disorder, hypersplenism (diagnosed by splenomegaly noted by palpation or ultrasonography, cytopenia, and hematopoietic cell hyperplasia in the bone marrow)；
13. The equivalent dose of corticosteroids used cumulatively within 7 days prior to apheresis was ≥ 70 mg prednisone；
14. Concomitant anticancer drugs or therapies (including radiotherapy);
15. Occurrence of a stroke or epileptic seizure within 6 months prior to signing the ICF;
16. Administration of live attenuated vaccine within 4 weeks prior to apheresis;
17. Major surgery within 2 weeks prior to apheresis, or scheduled surgery during the study or within 2 weeks after administration of study treatment. (Note: Subjects who plan to undergo surgery under local anesthesia may participate in the study.)
18. Any condition that is not conducive to the subject's ability to receive or tolerate the planned treatment at the study site, or understand the informed consent form, or any condition that, in the opinion of the investigator, is not in the best interest of the subject (e.g., impairing health), or any condition that may prevent, limit, or confound protocol-specified assessments.
19. Known life threatening allergic reactions, hypersensitivity reactions, or intolerance to LCAR-L10D cell formulation or their excipients, including DMSO (see Investigator's Brochure).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Type, incidence and severity of dose-limiting toxicities (DLTs) and treatment-emergent adverse events (TEAEs) | Day 1-90 days after injection
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose. An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment
Chimeric Antigen Receptor T（CAR-T）Positive Cell Concentration | Day 1-90 days after injection
  Venous blood samples will be collected for measurement of CAR-T positive cellular concentration

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) of this cell therapy | Day 1-90 days after injection
  Recommended Phase 2 dose (RP2D)
Overall response rate (ORR) after administration | 2 years post infusion
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LCAR-L10Dcell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per Lugano 2014 only.
Duration of remission (DOR) after administration | 2 years post infusion
  Duration of Remission (DOR) is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to LUGANO 2014 ) of the responders (who achieve PR or better response).
Progress Free Survival (PFS) after administration | 2 years post infusion
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LCAR-L10Dto the first documented disease progression (according to LUGANO 2014 ) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | 2 years post infusion
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-L10Dto death of the subject.
Time to Response (TTR) after administration | 2 years post infusion
  Time to Response (TTR) is defined as the time from the date of first infusion of LCAR-L10Dto the date of the first response evaluation of the subject who has met all criteria for PR or better.
Incidence of anti-LCAR-L10D antibody and positive sample titer | Day 1-90 days after injection
  Venous blood samples will be collected to measure LCAR-L10Dpositive cell concentrations and the transgenic level of LCAR-L10D, at the time points when anti-LCAR-L10D antibody serum samples are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aili He, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided